CLINICAL TRIAL: NCT06107686
Title: A Multicenter, Open-Label, Phase II Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of YL202 in Selected Patients With Advanced Solid Tumors
Brief Title: A Study of YL202 in Selected Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL202-CN-201-01
Record Dates: First submitted 2023-10-20; First posted 2023-10-30 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: NSCLC; Breast Cancer; HNSCC; Locally Advanced or Metastatic Solid Tumors
Keywords: Antibody-drug conjugate
MeSH Terms: conditions — Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Corhort A (Experimental): YL202 is provided as the lyophilized powder, 200 mg/vial. Locally advanced or metastatic NSCLC patients will be given YL202 by intravenously once every 3 weeks (Q3W) as a cycle.
  Interventions: Drug: YL202 should be intravenously infused
- Corhort B (Experimental): YL202 is provided as the lyophilized powder, 200 mg/vial. Locally advanced or metastatic BC patients will be given YL202 by intravenously once every 3 weeks (Q3W) as a cycle.
  Interventions: Drug: YL202 should be intravenously infused
- Corhort C (Experimental): YL202 is provided as the lyophilized powder, 200 mg/vial. Locally advanced or metastatic HNSCC patients will be given YL202 by intravenously once every 3 weeks (Q3W) as a cycle.
  Interventions: Drug: YL202 should be intravenously infused
- Corhort D (Experimental): YL202 is provided as the lyophilized powder, 200 mg/vial. Other locally advanced cancer patients will be given YL202 by intravenously once every 3 weeks (Q3W) as a cycle.
  Interventions: Drug: YL202 should be intravenously infused

INTERVENTIONS:
Drug: YL202 should be intravenously infused — For each patient, YL202 should be intravenously infused over 60±10 min.

SUMMARY:
This study is a multicenter, open-label, phase II study of YL202 in China to evaluate the efficacy, safety, and PK characteristics of YL202 in the following selected patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, phase II study of YL202 in China to evaluate the efficacy, safety, and PK characteristics of YL202 in the advanced NSCLC/BC/HNSCC/colorectal cancer/HER2-positive gastric cancer/cervical cancer/ovarian cancer and etc.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are aware of relevant trial information before the start of the trial, and voluntarily sign and date on the informed consent form (ICF).
2. Subjects aged from 18-75 (inclusive) years.
3. Histologically or cytologically confirmed at diagnosis of NSCLC/BC/HNSCC/other locally advanced or metastatic solid tumors including but not limited to colorectal cancer, HER2-positive gastric cancer, cervical cancer, ovarian cancer, etc..
4. At least one extracranial measurable lesion according to RECIST 1.1.
5. Archived or fresh tumor tissue samples can be provided.
6. With Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
7. The function of organs and bone marrow meets the requirements within 7 days before the first dose.
8. Female subjects of childbearing potential must agree to adopt highly effective contraceptive measures from screening throughout the study period and within at least 6 months after the last dose of the investigational product. Male subjects must agree to adopt highly effective contraceptive measures from screening throughout the study period and within at least 6 months after the last dose of the investigational product.
9. With expected survival ≥ 3 months.
10. Be capable of and willing to comply with the visits and procedures stipulated in the study protocol.

Exclusion Criteria:

1. With prior drug therapy targeting HER3 (including antibodies, antibody-drug conjugates [ADCs]), chimeric antigen receptor T-cell immunotherapy (CAR-T), and other drugs).
2. Previously intolerant to topoisomerase I inhibitors or ADC therapy composed of topoisomerase I inhibitors.
3. Are participating in another clinical study, unless it is an observational (non-interventional) clinical study or in the follow-up period of an interventional study.
4. The washout period from the previous anti-tumor therapy is insufficient before the first dose of the investigational product.
5. Patients who have received major surgery (excluding diagnostic surgery) within 4 weeks before the first dose of the investigational product or those who are expected to receive major surgery during the study.
6. Prior treatment with allogeneic bone marrow transplantation or solid organ transplantation.
7. Prior treatment with systemic steroids (prednisone > 10 mg/day or equivalent) or other immunosuppressive treatment within 2 weeks before the first dose of the investigational product.
8. Patients who have received any live vaccine within 4 weeks before the first dose of the investigational product or those who plan to receive live vaccine during the study period.
9. With meningeal metastasis or cancerous meningitis.
10. With brain metastasis or spinal cord compression.
11. Patients with uncontrolled or clinically significant cardiovascular diseases.
12. Clinically significant complicated pulmonary disorders.
13. Patients diagnosed with Gilbert syndrome.
14. Those with uncontrolled effusion in the third space requiring repeated drainage.
15. With a medical history of gastrointestinal perforation and/or fistula within 6 months before the first dose, or with active gastric and duodenal ulcers, ulcerative colitis, or other gastrointestinal diseases that may lead to hemorrhage or perforation according to the investigator.
16. With serious infection before the first dose.
17. With known human immunodeficiency virus (HIV) infection.
18. With active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
19. With a medical history of any other primary malignancies within 5 years before the first dose of the investigational product.
20. Unrelieved toxicity of previous anti-tumor therapy.
21. With a history of severe hypersensitivity to inactive ingredients in the raw materials and drug product or other monoclonal antibodies.
22. Lactating women, or women who are confirmed pregnant via a pregnancy test within 3 days before the first dose.
23. With any diseases, medical conditions, organ system dysfunction, or social conditions that may interfere with the ability of subjects to sign the ICF, adversely affect the ability of subjects to cooperate and participate in the study, or affect the interpretation of study results, including but not limited to mental illness or substance/alcohol abuse, in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
ORR assessed according to RECIST v1.1 | By the end of trial date, approximately within 36 months
  ORR: defined as the proportion of patients who achieved a best overall response of complete response (CR) or partial response (PR).
Determination of the recommended dose of YL202 in the pivotal clinical study | By the end of trial date, approximately within 36 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) assessed according to RECIST v1.1 | approximately within 36 months
Clinical benefit rate (CBR) assessed according to RECIST v1.1 | approximately within 36 months
depth of response (DpR) assessed according to RECIST v1.1 | Approximately within 36 months
disease control rate (DCR) assessed according to RECIST v1.1 | Approximately within 36 months
duration of response (DOR) assessed according to RECIST v1.1 | Approximately within 36 months
time to response (TTR) assessed according to RECIST v1.1 | Approximately within 36 months
Evaluate the overall survival (OS) | Approximately within 36 months
Adverse event (AE), described in terms of type, frequency, severity, time, and relationship with study treatment | Approximately within 36 months
Characterize the PK parameter AUC | Approximately within 36 months
  steady-state area under curve (AUC)
Characterize the PK parameter Cmax | Approximately within 36 months
  peak concentration (Cmax)
Characterize the PK parameter Ctrough | Approximately within 36 months
  trough concentration (Ctrough)
Characterize the PK parameter CL | Approximately within 36 months
  clearance (CL)
Characterize the PK parameter Vd | Approximately within 36 months
  volume of distribution (Vd)
Characterize the PK parameter t1/2 | Approximately within 36 months
  half-life (t1/2)
Incidence of anti-YL202 antibody | approximately within 36 months
Establish a POP PK model for exposure-response relationship analysis | approximately within 36 months
Evaluate the relatonship between different levels of HER3 expression and the sum of CR rate, PR rate and SD rate | approximately within 36 months

CONTACTS AND LOCATIONS:
Locations (80):
- China (80):
  - Anhui Tumour Hospital, Hefei, Anhui
  - The first affiliated hospital of Anhui Medical University, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chinese First Affiliated Hospital of Army Medical University of the People's Liberation Army, Chongqing, Chongqing Municipality
  - Chongqing University Affiliated Tumor Hospital, Chongqing, Chongqing Municipality
  - The first affiliated hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Xinqiao Hospital of AMU, Chongqing, Chongqing Municipality
  - Xinqiao Hospital, Chongqing, Chongqing Municipality
  - Fujian Tumor Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Shantou University Medical College Tumour Hospital, Shantou, Guangdong
  - Guilin Medical College Second Affiliated Hospital, Guilin, Guangxi
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Guangxi Medical University Affiliated Tumour Hospital, Nanning, Guangxi
  - The People's Hospital of Guangxi, Nanning, Guangxi
  - Harbin Medical university cancer hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital Of Henan University&Technology, Luoyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Xinxiang Medical University No.1 Affiliated Hospital, Xinxiang, Henan
  - He'nan Cancer Hospital South Gate, Zhengzhou, Henan
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Peoples Hospital of Jingzhou, Jingzhou, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - Union Hospital Tongji Medical College HuaZhong University of Science Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hu'nan Province Cancer Hospital, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya hospital Central South University, Changsha, Hunan
  - The Third People's Hospital of Hunan Province, Yueyang, Hunan
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Jilin Provincial Cancer Hospital, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The second Hospital of Dalian Medical University, Dalian, Liaoning
  - Fukuang General Hospital of Liaoning Health Industry Group, Fushun, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University Physical Examination Center, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong
  - Shandong Provincial Public Health Clinical Center, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Linyi Cancer hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The Affiliated Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The No.10 Peoples Hospital, Shanghai, Shanghai Municipality
  - Shanxi Province Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital Of Xi'an JiaoTong University, Xian, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - SiChuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - West China Hospital,Sichuan Universtiy, Chengdu, Sichuan
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Tumor Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University school of Medicine, Hangzhou, Zhejiang
  - ZheJiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Province People's Hospital, Hangzhou, Zhejiang
  - Zhejiang University Medical College Affiliated No.1 Hospital, Hangzhou, Zhejiang
  - Yiwu Central Hospital, Jinhua, Zhejiang
  - Taizhou Hospital of Zhejiang, Taizhou, Zhejiang